CLINICAL TRIAL: NCT06534203
Title: An Investigation of the Physical Task Demands of Caregivers Working in a Long-Term Care Facility in New Brunswick
Brief Title: Physical Task Demands of Caregivers Working in a Long-Term Care Facility
Status: Recruiting | Type: Observational
Sponsor: Universite de Moncton (Other)
Collaborators: University of New Brunswick (Other)
Responsible Party: Principal Investigator, Michelle Cardoso, Assistant Professor, Universite de Moncton
Other Study IDs: UMoncton
Record Dates: First submitted 2024-06-03; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Work Related Musculoskeletal Injuries (WRMSIs)
Keywords: Musculoskeletal Injuries; Healthcare; Patient Handling; Nursing Homes; Injury Prevention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Investigation - Observational Study — In this study, there will be no intervention, instead, it will be an observational study aimed at identifying the specific physical demands of caregivers working in long-term care facilities. This information will inform future interventions that can help reduce the occurrence of work-related musculoskeletal injuries.

SUMMARY:
Providing care to residents and patients significantly contributes to work-related injuries among healthcare personnel, particularly those responsible for transferring and handling residents, who face a higher risk of injury due to the physical demands of their work and other environmental factors.

The purpose of this project is to better understand the daily work requirements, identify their physical demands, and assess injury risk of caregivers. Data will be collected using a new pen-and-paper-based ergonomic surveying tool, a series of questionnaires, and measurements of physiological demands such as heart rate and galvanic skin response.

Collecting this data will enable the investigators and others to create new interventions better tailored to this working population, with a focus on injury prevention. These interventions may include warm-up routines, stretching exercises, training programs, and/or technological advancements.

DETAILED DESCRIPTION:
Purposes/Objectives:

The overall aim of this study is to establish a database on the physical requirements of caregivers working in long-term care homes.

This study will highlight the support needed for caregivers in long term care facilities, aiming to improve their working conditions through interventions and strategies that ensure their physical and mental well-being.

Research Questions:

The research question for this study is as follows:

1. What are the physical/musculoskeletal demands and motor movement patterns performed by caregivers in residential settings, and what does a typical workday entail for this population?
2. Is there a significant increase in perceived discomfort levels among caregivers throughout their workday?
3. What are the lifestyle habits of caregivers, and what is the prevalence and history of musculoskeletal injuries among caregivers?
4. Is there an increase in the fluctuations of their stress levels and heart rate throughout their workday?

Hypotheses:

The hypotheses for this study are as follows:

1. Caregivers spend a significant portion of their workday transferring residents or engaging in various repetitive motor tasks.
2. Caregivers experience significant increases in perceived discomfort in most areas of the body, which will be exacerbated throughout their shift.
3. There will be a correlation between lifestyle habits and injury history among caregivers.
4. Physiological stress levels will increase over the course of a caregiver's workday.

Introduction:

One of the key objectives of this study is to identify the physical demands and requirements of caregivers working in long-term care facilities. The first step involved creating an ergonomic tool tailored to the assessment of caregivers (See appendix A). This tool enables the recording of various motor tasks, behaviors and habits performed repetitively during a typical workday. Additionally, it facilitates the quantification of data to gain a better understanding of the physical demands of their work. This tool will allow investigators to determine the total time spent on specific motor tasks during a workday for this population.

In conjunction with the ergonomic tool, the investigators will administer questionnaires to gather information on lifestyle habits, work-related injury history, perceptions of job-related physical demands (using the Health and Lifestyle Questionnaire), and levels of discomfort during a workday (using the Rate of Perceived Discomfort Questionnaire (RPD-Q)). Additionally, physiological changes, such as galvanic skin response and heart rate fluctuations, will be recorded during data collection to monitor caregivers' physiological responses throughout the workday. This research approach will provide a comprehensive overview of the physical demands and injury risks amongst caregivers working in a long-term care facility. Collecting this data, will enable researchers and others in creating new interventions better tailored to this working population, such as warm-up routines, stretching exercises, training programs and/or technological advancements.

Methods:

This study employs mixed methods research, gathering both quantitative and qualitative data to comprehensively understand the issues surrounding Work Related Musculoskeletal Injuries (WRMSI) among caregivers in long-term care facilities in New Brunswick.

30 full-time caregivers from the York Care Center Nursing Home in Fredericton, Kenneth E Spencer Memorial Nursing Home in Moncton and Westford Nursing Home in Port Elgin will be recruited for this research project.

The participants will be caregivers working with residents with a level three classification. This means that the residents require constant supervision, may or may not be living with a stable chronic condition, and require assistance with personal care, sanitation, and mobility. All participants will be assessed for an 8 to 12-hour workday in a single experimental session.

The equipment used in this study includes:

1. A newly developed Pen-and-Paper based Ergonomic monitoring tool, designed by the researchers to identify the physical demands of caregivers' work, will be utilized in this study (see appendix A). The main objective of this research is to identify the different motor tasks, transfer procedures, positions and behaviors that pose risks of developing WRMSI in caregivers. The researchers will monitor and manually input each task performed by the caregivers.
2. The Rate of Perceived Discomfort Questionnaire (RPD-Q) (see appendix B) will be administered to track the progression of caregivers' discomfort during their workday. The RPD-Q is a self-reported questionnaire with a 100-point visual analogue scale that indicates the level of discomfort relative to specific body parts. A scale of point 0 corresponds to no discomfort and point 100 represents the worst discomfort imaginable; each point is the equivalent of one millimeter. Twenty-four different body parts will be measured in the RPD questionnaire on both the right and left sides of the body. The RPD questionnaire will be administered 3 times throughout the shift: Prior to the start of the shift, at the midpoint, and at the end of the caregiver's workday. Recording the RPD questionnaire at these specific timepoints will provide a snapshot on how discomfort levels develop throughout a typical working shift.
3. A questionnaire on lifestyle habits and work-related injury history (see appendix C) will be administered during data collection to gain insights into current lifestyle and previous workplace injury history of participants. The questionnaire is composed of short-answer, multiple-choice and open-ended questions that can be used as a journal during data collection. The H&L questionnaire will be filled out once during the workday of data collection. The objective of this questionnaire is to further understand the relationship between current lifestyle of the workers and the development of workplace injuries. The questionnaire is divided into three different subsections:

   * The amount of time spent in sedentary behavior, the amount of physical activity performed, and the amount of alcohol and tobacco consumed by participants in a typical week.
   * The number of years of experience in the sector, and participants' subjective perception of the physical demands imposed by their work.
   * The occurrence or non-occurrence of persistent work-related musculoskeletal injuries or discomfort, and the limitations these injuries impose on individuals' ability to work and their overall well-being.
4. Physiological Measures: An Empatica EmbracePlus watch, a galvanic skin response system, will be used to assess and quantify the participants' stress levels throughout their workday. Additionally, the Polar H10 heart rate monitor will enable the observation of caregivers' heart rate fluctuations during their workday. Data collection will follow a baseline measurement of participants heart rate and stress level, which will be taken after 5 minutes in a seated position, in a quiet area and with eyes closed prior to the start of their shift. Field notes will also be taken to facilitate the identification of the periods of the day when physiological stress levels are highest during data collection.

Statistical Analysis/Data Processing:

Descriptive Statistics:

Descriptive statistics using the software IMB SPSS, Version 29 (mean, median, standard deviation, etc.) will be used to evaluate quantitative values derived from the newly developed ergonomic tool.

Cross Correlations:

A series of cross correlations will be run on the Health and Lifestyle Questionnaire to identify correlations between different Work-Related Musculoskeletal Injury (WRMSI) risk factors. The correlation coefficient will enable the investigators to identify whether the relationships are inversely proportional or directly proportional. For example, it will be possible to examine the correlation between physical activity levels and WRMSI history, as well as whether there is a relationship between increases in smoking and alcohol consumption and WRMSI.

Repeated Measures ANOVA:

A Repeated Measure ANOVA will be used to interpret the results obtained from the RPD-Q. The data will be compared at three different time points: the beginning, middle and end of the caregiver's shift. During analysis, it will be possible to observe whether there has been a significant increase in perceived discomfort during the workday and which areas of the body experienced the most significant increase. Prior to running the repeated measures ANOVA, each data point will be plotted to observe if it is normally distributed. Mauchly's test will be used to assess the sphericity assumption. If the sphericity assumption is violated, the Greenhouse-Geisser correction will be used. The alpha level will be set at p < .05, and if any significant interactions are found, Tukey and Bonferroni post hoc analyses will be used.

The same approach will be used for the physiological outcome measures: heart rate monitor and the galvanic skin response system. Repeated Measures ANOVA will be utilized to compare the data collected at the beginning, middle and end of the caregiver's shift. The outcome measure will be to quantify whether stress levels and fluctuations of heart rate increased throughout the workday. If any significance is found, a Tukey and Bonferroni correction will be applied.

Qualitative Results:

A qualitative approach will be used to synthesize information gathered from the workers through the use of field notes. This will include documenting the circumstances surrounding their previous injuries and other relevant details.

ELIGIBILITY:
Inclusion Criteria:

* Full-time caregivers
* Caregivers responsible for the care and handling of residents
* Aged 19 or over

Exclusion Criteria:

* Part-time caregivers
* Caregivers not responsible for residents care and handling
* Caregivers under 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Full time caregivers working in a long term care facility responsable of resident care in New-Brunswick, Canada
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pen and Paper Ergonomic Tool - Part 1A : "The caregiver did NOT use any tools or aids while performing the following transfer tasks" | One experimental session (8 to 12 hours)
  Each participant will be observed throughout an entire workday using a new pen-and-paper-based ergonomic tool developed in the lab. This assessment tool (see Appendix A) is a comprehensive document designed to record the various physical tasks and demands encountered during a typical workday for caregivers in long-term care facilities. The tool was developed based on standardized task analysis tools widely used in ergonomic practices (OHCOW, 2023).
  Part 1A of this tool will identify the number of transfers performed by caregivers during a workday, specifying the frequency (number of times this task was performed) and time (seconds) of each type of transfer WITHOUT the use of tools or aids.
Pen and Paper Ergonomic Tool - Part 1B : "The caregiver used tools and/or aids while performing the following transfer tasks" | One experimental session (8 to 12 hours)
  Part 1B of this tool will identify the number of transfers performed by caregivers during a workday, specifying the frequency (number of times this task was performed) and time (seconds) for each type of transfer WITH the use of tools or aids.
Pen and Paper Ergonomic Tool - Part 1C: "Tools used for resident transfers" | One experimental session (8 to 12 hours)
  The purpose of Part 1C is to determine how many transfers each type of equipment was used for by caregivers on a workday. It identifies the frequency of use for both mechanical and non-mechanical tools.
Pen and Paper Ergonomic Tool - Part 2A: "Number of resident handling in Bed" | One experimental session (8 to 12 hours)
  Part 2A of this tool will identify the number of resident handling tasks performed by caregivers in bed during a workday, specifying the frequency (i.e., the number of times this task was performed). This section is also subdivided to identify not only the number of manipulations but also the types of manipulations performed.
Pen and Paper Ergonomic Tool - Part 2B: "Number of resident handling in Wheelchair - Sitting" | One experimental session (8 to 12 hours)
  Part 2B of this tool will identify the number of resident handling tasks performed by caregivers in a wheelchair or sitting position during a workday, specifying the frequency (i.e., the number of times this task was performed). This section is also subdivided to identify not only the number of manipulations but also the types of manipulations performed.
Pen and Paper Ergonomic Tool - Part 3: "Motor tasks - Housework - Sanitary" | One experimental session (8 to 12 hours)
  Sanitary services and needs, such as bending down to clean or pick up objects, can expose caregivers to risks of WRMSIs, especially if they are in a vulnerable position while performing motor tasks. Assisting residents with hygiene care and clothing changes can also vary in terms of time and complexity, which can present challenges for caregivers and increase their risk of injury. This section of the tool will provide an overview of the frequency with which these types of motor tasks are performed during a workday.
Pen and Paper Ergonomic Tool - Part 4: "Time spent under different type of behavior" | One experimental session (8 to 12 hours)
  Extended periods of standing and walking can have significant long-term effects on health. Therefore, this section is crucial as it allows for the recording of the approximate time (in minutes) spent on various activities, such as standing, sitting, and walking, throughout a workday.
Pen and Paper Ergonomic Tool - Part 5: "Additional information" | One experimental session (8 to 12 hours)
  This section of the tool will identify several important factors that can influence the risk of injury to caregivers, including the total time worked during the shift, rest periods, and the longest continuous period worked without rest (in minutes).
Pen and Paper Ergonomic Tool - Part 6: "Field observations" | One experimental session (8 to 12 hours)
  This section of the tool will be used to record any additional behaviors, factors, or obstacles that may increase the risk of injury to caregivers and that have not been covered elsewhere in the tool. It will serve as a journal for the investigators to track valuable information during data collection.

SECONDARY OUTCOMES:
Rate of Perceived Discomfort Questionnaire (RPD-Q) | One experimental session (8 to 12 hours)
  The RPD-Q will be administered to provide an overview of the progression of caregivers' discomfort during their workday. This questionnaire will quantify the discomfort felt by the participants at the beginning, during, and after their workday during data collection. This self-administered questionnaire is based on a visual analogue scale of 0 to 100 points. Zero points represent no discomfort at all, while 100 points represent the maximal level of discomfort. Additionally, the RPD-Q will make it possible to identify whether the level of discomfort increases as the workday progresses, as well as the areas of the body most affected by such changes.

OTHER OUTCOMES:
Health and Lifestyle Questionnaire - Part 1A : "Lifestyle Habits" | One experimental session (8 to 12 hours)
  To gain an overview of work-related injuries in a care setting, investigators will gather information to identify risk factors and determine whether certain habits might contribute to injury development within this population. The H&L-Q is divided into three parts, with the first focusing on lifestyle habits, such as average alcohol consumption (in ounces) during a typical week.
Health and Lifestyle Questionnaire - Part 1B : "Lifestyle Habits" | One experimental session (8 to 12 hours)
  This section of the questionnaire provides relevant information regarding lifestyle habits, such as average tobacco use during a typical week. The outcome measurement will be based on the frequency of use throughout the week.
Health and Lifestyle Questionnaire - Part 1C : "Lifestyle Habits" | One experimental session (8 to 12 hours)
  This section of the questionnaire provides relevant information regarding lifestyle habits, including the estimated amount of time engaging in physical activities (in minutes) and time spent in sedentary behavior (in hours) during a week.
Health and Lifestyle Questionnaire - Part 2 : "Work related MSIs History" | One experimental session (8 to 12 hours)
  This section captures the history of WRMSIs experienced by participants throughout their careers. It aims to assess the impact of these injuries on their work capacity and overall well-being. By analyzing this data, investigators will be able to determine the prevalence of WRMSIs (%) within the study population.
Health and Lifestyle Questionnaire - Part 3 : "Subjective Information" | One experimental session (8 to 12 hours)
  This section includes subjective data from participants to aid in interpreting results obtained from other tools. It also features open-ended questions designed to gather insights on interventions and strategies that could help reduce the occurrence of WRMSIs among caregivers.
Physiological Measures - Galvanic Skin Response Levels | One experimental session (8 to 12 hours)
  The use of an Empatica (Embrace Plus) watch will allow investigators to assess the physiological demands placed on caregivers throughout their workday. By monitoring fluctuations in galvanic skin response levels, researchers can quantify physiological responses and identify the most stressful periods of a shift by analyzing electrical conductance in microsiemens (µS).
Physiological Measures - Heart Rate | One experimental session (8 to 12 hours)
  The use of the heart rate monitor (Polar H10) will enable investigators to assess the physiological demands on caregivers throughout their workday. By analyzing fluctuations in heart rate (beats per minute, bpm), it will be possible to identify the more physically demanding periods of a caregiver's shift. Additionally, the average heart rate throughout the workday can be calculated to quantify the overall physical demands imposed on caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cardoso, PhD, Principal Investigator — Université de Moncton; Wayne Albert, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- Université de Moncton, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT06534203/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT06534203/SAP_001.pdf
  • Informed Consent Form (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT06534203/ICF_002.pdf